CLINICAL TRIAL: NCT04684394
Title: A Multicenter, Multiple-Dose Study in Neovascular Age-related Macular Degeneration (nAMD) to Evaluate the Safety, Tolerability, Pharmacodynamics, Immunogenicity, and Clinical Effect of Repeat Intravitreal (IVT) Injections of GEM103 as an Adjunct to Standard of Care Aflibercept Therapy
Brief Title: A Multiple Dose Study of Repeat Intravitreal Injections of GEM103 in Neovascular Age-related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Gemini Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEM-CL-10311
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-03

CONDITIONS: Neovascular Age-related Macular Degeneration; Retinal Disease; Retinal Degeneration; Macular Degeneration
MeSH Terms: conditions — Retinal Diseases; Retinal Degeneration; Macular Degeneration | interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SoC + GEM103 (Experimental): Participants were administered SoC therapy defined as aflibercept (2 milligram [mg]/50 microliter [mcL]) first, followed by GEM103 (500 microgram [mcg]/50mcL) 15 minutes later. Administration occurred every other month (EOM) for a total of 6 doses during the 12-month study period.
  Interventions: Biological: GEM103; Drug: Aflibercept
- SoC + Sham (Sham Comparator): Participants were administered SoC therapy defined as aflibercept (2mg/50mcL) first, followed by the Sham injection 15 minutes later. Administration occurred EOM for a total of 6 doses during the 12-month study period.
  Interventions: Drug: Aflibercept; Drug: Sham

INTERVENTIONS:
Biological: GEM103 — GEM103 500 mcg/50 mcL intravitreal injection
  Arms: SoC + GEM103
Drug: Aflibercept — Aflibercept 2 mg/50 mcL (SOC) intravitreal injection
  Sham intravitreal injection
Drug: Sham — Sham intravitreal injection
  Arms: SoC + Sham

SUMMARY:
This study is designed to investigate the safety and tolerability of GEM103 IVT injection + standard of care vs. sham + standard of care.

DETAILED DESCRIPTION:
This is a Phase 2a, multi-center, multiple dose study in subjects with Neovascular Age-related Macular Degeneration (nAMD) to investigate the safety and tolerability of GEM103 IVT injection + standard of care vs. sham + standard of care.

Subjects will undergo clinical and ophthalmic assessments for determination of inclusion in the study and who meet all eligibility criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. At least 50 years old at the time of signed informed consent
2. Choroidal neovascularization (CNV) related to nAMD with the following features, as determined by the Image Reading Center

   1. Maximum CNV lesion size of 12 disc areas
   2. Subretinal hemorrhage less than or equal to (<=) 50% of lesion size
3. On aflibercept treatment prior to Day 1
4. Best Corrected Visual Acuity (BCVA) in the study eye between 24 to 75 letters using EDTRS

Exclusion Criteria:

1. Presence of the following ocular conditions in the study eye:

   1. Any active ocular disease or condition that impact the subject to participate in the study or be a contraindication of IVT injections
   2. Any intraocular surgery
   3. Aphakia or complete absence of the posterior capsule
   4. Prior corneal transplant
   5. Scar or fibrosis greater than or equal to (>=) 50% of CNV lesion or involving center of fovea
2. Presence of any of the following ocular conditions in either eye:

   1. History of herpetic infection, idiopathic polypoidal choroidal vasculopathy (PCV), pathologic myopia, central serous chorioretinopathy (CSCR), adult onset foveal pattern dystrophy
   2. Concurrent disease that could require medical or surgical intervention during the study period
   3. Active/suspected ocular/periocular infection or active intraocular inflammation
   4. History of idiopathic or autoimmune-associated uveitis
3. Any prior or ongoing medical condition or clinically significant screening laboratory value that may present a safety risk, interfere with study compliance, interfere with consistent study follow-up, or confound data interpretation throughout the longitudinal follow-up period
4. Has experienced a cardiovascular or cerebrovascular event within 12 months of informed consent
5. Females must not be pregnant or lactating
6. Current use of medications known to be toxic to the lens, retina or optic nerve
7. Use of any investigational new drug or other experimental treatment in the last 6 months prior to Day 1, and/or receipt of any prior gene therapy or ocular device implantation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Gemini Clinical Trial Site 16, Phoenix, Arizona
  - Gemini Clinical Trial Site 11, Campbell, California
  - Gemini Clinical Trial Site 9, Encino, California
  - Gemini Clinical Trial Site 17, Huntington Beach, California
  - Gemini Clinical Trial Site 12, Pasadena, California
  - Gemini Clinical Trial Site 5, Miami, Florida
  - Gemini Clinical Trial Site 7, Pinellas Park, Florida
  - Gemini Clinical Trial Site 20, Sarasota, Florida
  - Gemini Clinical Trial Site 8, Stuart, Florida
  - Gemini Clinical Trial Site 18, Winter Haven, Florida
  - Gemini Clinical Trial Site 19, Indianapolis, Indiana
  - Gemini Clinical Trial Site 4, Hagerstown, Maryland
  - Gemini Clinical Trial Site 23, Worcester, Massachusetts
  - Gemini Clinical Trial Site 22, Royal Oak, Michigan
  - Gemini Clinical Trial Site 1, Reno, Nevada
  - Gemini Clinical Trial Site 2, Asheville, North Carolina
  - Gemini Clinical Trial Site 15, Charlotte, North Carolina
  - Gemini Clinical Trial Site 6, Cincinnati, Ohio
  - Gemini Clinical Trial Site 10, Eugene, Oregon
  - Gemini Clinical Trial Site 13, Beaufort, South Carolina
  - Gemini Clinical Trial Site 3, Dallas, Texas
  - Gemini Clinical Trial Site 21, San Antonio, Texas
  - Gemini Clinical Trial Site 14, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at multiple sites in the United States from 29 December 2020 to 18 February 2022.
Pre-assignment Details: A total of 70 participants were screened of which 20 were screen failure. 50 participants were randomized in 2:1 ratio in this study, of which 34 participants received the GEM103 + aflibercept (SoC) and 16 received the Sham + SoC.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | SoC + GEM103 | SoC + Sham
Started | 34; 68 eyes | 16; 32 eyes
Study Eye | 34; 34 eyes | 16; 16 eyes
Fellow Eye | 34; 34 eyes | 16; 16 eyes
Completed | 5; 10 eyes | 1; 2 eyes
Not Completed | 29; 58 eyes | 15; 30 eyes
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Study discontinued per Sponsor decision | 25 | 13

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug (GEM103 or sham).
Groups:
- SoC + GEM103: Participants were administered SoC therapy defined as aflibercept (2mg/50mcL) first, followed by GEM103 (500mcg/50mcL) 15 minutes later. Administration occurred EOM for a total of 6 doses during the 12-month study period.
- Total: Total of all reporting groups
Arm/Group | SoC + GEM103 | SoC + Sham | Total
Number analyzed (Participants) | 34 | 16 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 34 | 16 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 11 | 31
  Male | 14 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 32 | 16 | 48
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 16 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence or worsening of a pre-existing condition in a participant administered a pharmaceutical product during the study, whether related or not to the study medication. TEAEs were defined as AE that occurred on or after the date and time of study drug administration or those that first occurred pre-dose but worsened by increase in occurrence or severity after study drug administration. Number of participants with ocular TEAEs in study eye and fellow eye were reported.
Time Frame: Baseline up to Week 48
Population: The FAS included all randomized participants who received at least 1 dose of study drug (GEM103 or sham).
Measure: Count of Participants; unit: Participants
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 34 | 16
Participants
  Participants with Ocular TEAE in Study Eye | 11 | 1
  Participants with Ocular TEAE in Fellow Eye | 6 | 3

2. Primary Outcome: Number of Participants With Non-ocular TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence or worsening of a pre-existing condition in a participant administered a pharmaceutical product during the study, whether related or not to the study medication. TEAEs were defined as AE that occurred on or after the date and time of study drug administration or those that first occurred pre-dose but worsened by increase in occurrence or severity after study drug administration. Number of participants with non-ocular TEAEs were reported.
Time Frame: Baseline up to Week 48
Population: The FAS included all randomized participants who received at least 1 dose of study drug (GEM103 or sham).
Measure: Count of Participants; unit: Participants
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 34 | 16
Participants | 10 | 7

3. Primary Outcome: Number of Participants With Abnormal Ophthalmic Examination Findings
Description: Ophthalmoscopy examination was performed in each eye with findings reported for Vitreous, Optic Nerve, Macula, Retina Periphery. Lens Status and Opacification (Phakic and Pseudophakic) was also performed. Nuclear Cataract, Cortical Cataract, and Posterior Subcapsular Cataract categories was further summarized by severity grade. Ocular biomicroscopic examination was performed with findings reported for Lids/Lashes, Conjunctiva, Cornea, Anterior Chamber, and Iris/Pupil.
Time Frame: Baseline up to Week 48
Population: The FAS included all participants who received at least 1 dose of study drug/reference therapy (GEM103 or sham). Here "overall number of participants analyzed" are those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 29 | 13
Participants
  Participants With Vitreous in Study Eye | 26 | 8
  Participants With Vitreous in Fellow Eye | 23 | 8
  Participants With Optic Nerve in Study Eye | 4 | 5
  Participants With Optic Nerve in Fellow Eye | 4 | 6
  Participants With Macula in Study Eye | 28 | 11
  Participants With Macula in Fellow Eye | 28 | 12
  Participants With Retina Periphery in Study Eye | 5 | 2
  Participants With Retina Periphery in Fellow Eye | 6 | 4
  Participants With Phakic in Study Eye | 5 | 4
  Participants With Phakic in Fellow Eye | 6 | 5
  Participants With Pseudophakic in Study Eye | 24 | 9
  Participants With Pseudophakic in Fellow Eye | 23 | 8
  Participants With Nuclear Cataract: Mild in Study Eye | 1 | 1
  Participants With Nuclear Cataract: Mild in Fellow Eye | 2 | 1
  Participants With Nuclear Cataract: Moderate in Study Eye | 1 | 3
  Participants With Nuclear Cataract: Moderate in Fellow Eye | 1 | 4
  Participants With Nuclear Cataract: Severe in Study Eye | 2 | 0
  Participants With Nuclear Cataract: Severe in Fellow Eye | 2 | 0
  Participants With Cortical Cataract: Mild in Study Eye | 1 | 0
  Participants With Cortical Cataract: Mild in Fellow Eye | 2 | 1
  Participants With Cortical Cataract: Moderate in Study Eye | 0 | 0
  Participants With Cortical Cataract: Moderate in Fellow Eye | 0 | 0
  Participants With Cortical Cataract: Severe in Study Eye | 0 | 0
  Participants With Cortical Cataract: Severe in Fellow Eye | 0 | 0
  Participants With Posterior Subcapsular Cataract: Mild in Study Eye | 0 | 0
  Participants With Posterior Subcapsular Cataract: Mild in Fellow Eye | 0 | 0
  Participants With Posterior Subcapsular Cataract: Moderate in Study Eye | 0 | 0
  Participants With Posterior Subcapsular Cataract: Moderate in Fellow Eye | 0 | 0
  Participants With Posterior Subcapsular Cataract: Severe in Study Eye | 0 | 0
  Participants With Posterior Subcapsular Cataract: Severe in Fellow Eye | 0 | 0
  Participants With Lids/Lashes findings in Study Eye | 4 | 2
  Participants With Lids/Lashes findings in Fellow Eye | 5 | 2
  Participants With Cornea findings in Study Eye | 8 | 3
  Participants With Cornea findings in Fellow Eye | 6 | 1
  Participants With Conjunctiva findings in Study Eye | 2 | 1
  Participants With Conjunctiva findings in Fellow Eye | 2 | 1
  Participants With Iris Pupil findings in Study Eye | 2 | 0
  Participants With Iris Pupil findings in Fellow Eye | 0 | 0
  Participants With Anterior Chamber findings in Study Eye | 1 | 0
  Participants With Anterior Chamber findings in Fellow Eye | 1 | 0

4. Primary Outcome: Percentage of Participants With Greater Than or Equal to (>=)15, >=10, >=5 Letters From the Baseline in Best Corrected Visual Acuity (BCVA)
Description: Visual function assessments included BCVA assessment in each eye by Early Treatment Diabetic Retinopathy Study (ETDRS) letters. BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The letter score ranges from 0 (worse score) to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average value was calculated across the three visits, and this averaged value was used to determine if the endpoint was met. The results were summarized as the percentage of participants with increase in BCVA with greater than or equal to (>=)15, >=10, >=5 letters from the baseline per treatment arm who met the endpoint.
Time Frame: Baseline up to Week 48
Population: The FAS included all randomized participants who received at least 1 dose of study drug (GEM103 or sham). Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 30 | 13
percentage of participants
  >=15 Letters in Study Eye | 0 | 0
  >=10 Letters in Study Eye | 3.3 | 0
  >=5 Letters in Study Eye | 43.3 | 15.4
  >=15 Letters in Fellow Eye | 3.3 | 7.7
  >=10 Letters in Fellow Eye | 6.7 | 15.4
  >=5 Letters in Fellow Eye | 23.3 | 15.4

5. Primary Outcome: Percentage of Participants With Greater Than or Equal to (>=)15, >=10, >=5 Letters From the Baseline in Low Luminance Visual Acuity (LLVA)
Description: Visual function assessments included LLVA assessment in each eye by ETDRS letters. LLVA was measured on the ETDRS chart at a starting distance of 4 meters. The letter score ranges from 0 (worse score) to 100 (best score), and a gain in LLVA from baseline indicates an improvement in visual acuity. For each participant, an average value was calculated across the three visits, and this averaged value was used to determine if the endpoint was met. The results were summarized as the percentage of participants with increase in LLVA with >=15, >=10, >=5 letters from the baseline per treatment arm who met the endpoint.
Time Frame: Baseline up to Week 48
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 30 | 13
percentage of participants
  >=15 Letters in Study Eye | 6.7 | 0
  >=10 Letters in Study Eye | 16.7 | 7.7
  >=5 Letters in Study Eye | 26.7 | 53.8
  >=15 Letters in Fellow Eye | 3.3 | 0.0
  >=10 Letters in Fellow Eye | 6.7 | 0.0
  >=5 Letters in Fellow Eye | 10.0 | 15.4

6. Primary Outcome: Mean Change From Baseline in Minnesota Low-vision Reading (MNRead) Test at Week 48
Description: The MNRead acuity cards are continuous-text reading acuity cards suitable for measuring the reading acuity and reading speed of normal and low-vision participants. Formula for reading speed words per minute (wpm): reading speed is equal to 60*(10 - errors)/ (time in seconds). A negative change from baseline indicates a decrease in the reading speed; disease worsening.
Time Frame: Baseline, Week 48
Population: The FAS included all randomized participants who received at least 1 dose of study drug (GEM103 or sham). Here, "overall number of participants analyzed, and overall number of units analyzed" signifies those participants and units respectively who were evaluable for this outcome measure and number of participants and units analyzed signifies those who were evaluable for specified categories.
Measure: Mean (Standard Error); unit: wpm
Units Other Than Participants: eyes
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 29 | 13
Number analyzed (eyes) | 58 | 26
wpm
  Study Eye: number analyzed (eyes) | 29 | 13
  Study Eye | -21.41 (7.070) | -30.35 (35.707)
  Fellow Eye: number analyzed (eyes) | 29 | 13
  Fellow Eye | -18.86 (63.209) | -7.88 (43.452)
  Both Eyes: number analyzed (Participants) | 28 | 13
  Both Eyes: number analyzed (eyes) | 56 | 26
  Both Eyes | -4.73 (47.397) | 3.08 (52.499)

7. Secondary Outcome: Change From Baseline in Total Complement Factor H (CFH) Concentration in Aqueous Humor
Description: Observed continuous total CFH concentration level in aqueous humor (ng/mL) was analyzed in study eye only by type of biological matrix by treatment group using descriptive statistics. Change from baseline in total CFH Concentration in aqueous humor at Week 32 was reported.
Time Frame: Baseline, Week 32
Population: The biomarker set (BS) included participants with sufficient data to assess biomarker results. Here, "overall number of participants analyzed, and overall number of units analyzed" signifies those participants and units respectively who were evaluable for this outcome measure and number of units analyzed signifies those who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Units Other Than Participants: eyes
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 1 | 1
Number analyzed (eyes) | 1 | 1
nanogram per milliliter (ng/mL) | 602.890 | 156.520

8. Secondary Outcome: Mean Change From Baseline in Early Treatment of Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) at Week 48
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters in each eye. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was used to determine if the endpoint was met. All items were transformed on to total score ranges from 0 to 100 (best score). A negative change indicates no improvement in the condition.
Time Frame: Baseline, Week 48
Population: The FAS included all randomized participants who received at least 1 dose of study drug (GEM103 or sham). Here, "overall number of participants analyzed, and overall number of units analyzed" signifies those participants and units respectively who were evaluable for this outcome measure and number of units analyzed signifies those who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 30 | 13
Number analyzed (eyes) | 60 | 26
ETDRS letters
  Study Eye: number analyzed (eyes) | 30 | 13
  Study Eye | 1.0 (8.44) | -0.4 (5.24)
  Fellow Eye: number analyzed (eyes) | 30 | 13
  Fellow Eye | 0.0 (11.05) | 0.7 (8.10)

9. Secondary Outcome: Mean Change From Baseline in Macular Atrophy (MA) Assessed by Fundus Autofluorescence (FAF)
Description: MA lesion area was measured in millimeters squared (mm^2) by FAF in each eye. The change in MA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of MA lesion area (worsening; disease progression).
Time Frame: Baseline up to Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimeters squared (mm^2)
Units Other Than Participants: eyes
Arm/Group | SoC + GEM103 | SoC + Sham
Number analyzed (Participants) | 1 | 0
Number analyzed (eyes) | 2 | 0
millimeters squared (mm^2)
  Study Eye: number analyzed (eyes) | 1 | 0
  Study Eye | 2.170 |
  Fellow Eye: number analyzed (eyes) | 1 | 0
  Fellow Eye | 2.430 |

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 48
Description: The FAS included all randomized participants who received at least 1 dose of study drug (GEM103 or sham). Overall data (Ocular and Non-Ocular) has been reported here.
Arm/Group | SoC + GEM103 | SoC + Sham
All-Cause Mortality (participants affected / at risk) | 1/34 | 2/16
Serious Adverse Events (participants affected / at risk) | 5/34 | 4/16
Other Adverse Events (participants affected / at risk) | 18/34 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SoC + GEM103 (N=34) | SoC + Sham (N=16)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SoC + GEM103 (N=34) | SoC + Sham (N=16)
Vitreous floaters (Eye disorders) | 3 | 0
Eye pain (Eye disorders) | 2 | 0
Retinal degeneration (Eye disorders) | 3 | 1
Vitreous detachment (Eye disorders) | 3 | 0
Cystitis (Infections and infestations) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Blood potassium increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Conjunctival deposit (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Macular degeneration (Eye disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Photopsia (Eye disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Punctate keratitis (Eye disorders) | 1 | 0
Retinal drusen (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 2 | 4
Retinopathy hypertensive (Eye disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Visual impairment (Eye disorders) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT04684394/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT04684394/SAP_001.pdf